CLINICAL TRIAL: NCT06684119
Title: Assessing Optimal Positive End-expiratory Pressure (PEEP) Using Electrical Impedance Tomography (EIT) During a PEEP Titration Protocol in Mechanically Ventilated Children with Pediatric Acute Respiratory Distress Syndrome (PARDS)
Brief Title: Pediatric Positive End Expiratory Pressure (PEEP) Titration Using Electrical Impedence Tomography (EIT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Anoopindar Bhalla, Medical Staff/USC Faculty, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-24-00295
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome
Keywords: positive end-expiratory pressure; Electrical Impedance Tomography; respiratory distress
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrical Impedance Tomography positive end-expiratory pressure (Experimental): Patients will be monitored using Electrical Impedance Tomography and the positive end-expiratory pressure titration tool as their positive end-expiratory pressure is adjusted according to a step wise positive end-expiratory pressure titration protocol.
  Interventions: Device: Electrical Impedance Tomography positive end-expiratory pressure titration

INTERVENTIONS:
Device: Electrical Impedance Tomography positive end-expiratory pressure titration — A PEEP titration will occur for the patient with the PEEP increased by 2 cm H2O every 2 minutes until a maximum PEEP of 20 or three steps (+ 6 cm H2O) above the set clinical PEEP. The PEEP will then be decreased by 2 cmH2O every 2 minutes until a minimum PEEP of 6 cmH2O or three steps (- 6 cm H2O) below their clinical PEEP.

SUMMARY:
The goal of this clinical trial is to perform a PEEP titration protocol and use EIT to identify the optimal PEEP at which lung overdistention and collapse are most effectively balanced. The primary and secondary aims of the study are as follows:

Identify the difference between the optimal PEEP recommended by EIT metrics and the current guideline recommended approach to identifying optimal PEEP in PARDS. There will be a statistically significant difference in the recommended optimal PEEP identified using the EIT PEEP titration tool and that of the PEEP/FiO2 grid recommendations.

Determine the difference in physiologic metrics between EIT optimal PEEP and the PEEP/FiO2 recommended PEEP.

Participants will undergoing EIT monitoring while being subjected to PEEP titration protocol.

ELIGIBILITY:
Inclusion Criteria:

* Any person who is less than 18 years of age
* is on invasive mechanical ventilation
* is not spontaneously breathing
* meets PARDS criteria

Exclusion Criteria:

* Contraindication to the use of EIT
* Hemodynamic instability
* Contraindications to hypercapnia
* patients with uncuffed endotracheal or tracheostomy tubes
* diagnosis of pneumothorax or bronchopleural fistula
* non-conventional ventilation
* any patient on extra-corporeal membrane oxygenation (ECMO) support
* less than 1 week post-operatively from cardiac surgery
* the following cardiac diagnoses: Glenn or Fontan physiology, significant right to left shunt
* Corrected Gestational Age < 37 weeks
* pregnancy

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The absolute difference between the electrical impedence tomography (EIT) recommended PEEP and the PEEP recommended by the PEEP/fraction of inspired oxygen (FiO2) grid. | Day 1
  Collected using electrical impedence tomography (EIT). The EIT device provides the percentages of alveolar overdistention and collapse at each PEEP level. The best PEEP by EIT is defined as the PEEP level above the intersection of curves representing relative alveolar overdistention and collapse.

SECONDARY OUTCOMES:
Lung recruitability, as measured by electrical impedence tomography, and its association with difference in optimal PEEP recommended by electrical impedence tomography versus the PEEP/FiO2 grid | Day 1
  Recruitability will be defined as the absolute reduction in the percentage of collapse when comparing the highest and lowest PEEP achieved, as measured by electrical impedence tomography.
Difference in systolic impendence, as a surrogate for cardiac output, using electrical impedence tomography at various PEEP levels | Day 1
  Using the electrical impedence tomography pulsatility filter/tool, a difference in systolic impendence, attributed to the cardiac cycle, can be calculated. This will be used as a surrogate for stroke volume and will be compared across PEEP levels.
Change in static compliance across different PEEP levels during a PEEP titration | Day 1
  Static compliance is defined as the change in volume divided by the change in pressure during an inspiratory hold (when airflow is zero). It reflects the elastic properties of the lung and chest wall.
Change in driving pressure across different PEEP levels during a PEEP titration | Day 1
  Driving pressure is the difference between the plateau pressure (the pressure measured during an inspiratory hold, when airflow is zero) and the positive end-expiratory pressure (PEEP). It represents the pressure that actually distends the alveoli during mechanical ventilation.
Change in plateau pressure across different PEEP levels during a PEEP titration | Day 1
  Plateau pressure is the pressure measured during an inspiratory hold maneuver, which occurs when the ventilator temporarily halts airflow at the end of the inspiratory phase. This allows the pressure in the alveoli to stabilize, providing a true reflection of the pressure needed to distend the lungs, without the effects of airflow resistance.
Change in dead space, as measured by volumetric capnography, across different PEEP levels during a PEEP titration | Day 1
  For patients who consent to the optional placement of a volumetric capnography device, dead space will be continuously measured using volumetric capnography by measuring the volume of carbon dioxide (CO2) exhaled with each breath (VeCO2) and calculating the CO2 ventilatory equivalent (minute ventilation/VCO2). Airway dead space can be obtained with each breath.
Change in transplural pressure, as measured by esophageal manometry, across different PEEP levels during a PEEP titration | Day 1
  For patients who consent to the optional component of having an esophageal balloon catheter placed, esophageal manometry will be used to measure transplural pressure. The difference between the pressure in the alveoli (intrapulmonary pressure) and the pressure in the pleural space (intrapleural pressure). It reflects the pressure required to expand the lungs and is crucial for understanding lung mechanics. This will be obtained using esophageal manometry with inspiratory and expiratory holds at each PEEP titration level.

CONTACTS AND LOCATIONS:
Overall Officials: Anoopindar Bhalla, MD, Study Director — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No